CLINICAL TRIAL: NCT02155725
Title: Study on the Efficacy and Safety of a Therapeutic Strategy of PPH Comparing Early Administration of Human Fibrinogen vs Placebo in Patients Treated With IV Prostaglandins Following Vaginal Delivery
Brief Title: Fibrinogen in Haemorrhage of Delivery
Acronym: FIDEL
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Laboratoire français de Fractionnement et de Biotechnologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIDEL; 2013-002484-26 (EudraCT Number)
Record Dates: First submitted 2014-05-20; First posted 2014-06-04 (Estimated); Results first posted 2020-09-25 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-07

CONDITIONS: Post-Partum Hemorrhage
Keywords: PPH; fibrinogen; vaginal delivery
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Human Fibrinogen concentrate (Experimental): 2 vials (200ml) / 3g intravenous
  Interventions: Drug: Human Fibrinogen concentrate
- Placebo (Placebo Comparator): 2 vials (200ml)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Human Fibrinogen concentrate — Injection as soon as possible and within 30 min following the start of prostaglandin infusion
  Other Names: Clottafact, LFB
  Arms: Human Fibrinogen concentrate
Drug: Placebo — As soon as possible and within 30 min following the start of prostaglandin infusion
  Arms: Placebo

SUMMARY:
The purpose of the study is to assess the benefits of a therapeutic strategy that associates an early administration of human fibrinogen concentrate in the management of PPH on the reduction of bleeding after the initiation of prostaglandins intravenous infusion, following vaginal delivery.

DETAILED DESCRIPTION:
Randomised, double-blind,multicenter, placebo-controlled study

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Vaginal delivery
* PPH requiring IV administration of prostaglandins
* At least one available result of Hb level during the third trimester of pregnancy
* 18-year-old female patients and older
* Covered by healthcare insurance in accordance with local requirements

Exclusion Criteria:

* Caesarean section
* Haemostatic intervention (as ligation, embolization or hysterectomy) already decided at the time of inclusion
* Known placenta praevia or accreta
* Hb level < 10g/dl during the third trimester of pregnancy
* History of venous or arterial thromboembolic event
* Known inherited bleeding or thrombotic disorders
* Treatment with low-molecular-weight heparin (LMWH) within 24 hours prior to the inclusion
* Treatment with acetylsalicylic acid within 5 days prior to the inclusion
* Treatment with vitamin K antagonists within 7 days prior to the inclusion
* Administration of fibrinogen concentrate within 48 hours prior to the inclusion
* Administration of FFP, platelets units or prohaemostatic drugs, tranexamic acid and rFVIIa or prothrombin complex concentrates (PCC) within 48 hours prior to the inclusion
* Administration of RBCs within 3 months prior to the inclusion
* Participation in another interventional clinical study within 30 days prior to the inclusion
* Previous inclusion/enrolment in the present clinical study
* Known history of hypersensitivity or other severe reaction to any component of Clottafact® or placebo
* Minors, majors under guardianship, persons staying in health or social institutes and people deprived of their freedom
* Known drug or alcohol abuse
* Patients whose use of concomitant medication may interfere with the interpretation of data
* Any other current significant medical condition that might interfere with treatment evaluation according to the investigator's judgement
* Patients who are unlikely to survive through the treatment period and evaluation
* Patients transferred from another service

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 448 (Actual)
Dates: Start 2014-04-10; Primary Completion 2018-08-06 (Actual); Study Completion 2018-08-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Sophie DUCLOY-BOUTHORS, Dr, Principal Investigator — Maternité Jeanne de Flandre - 59037 LILLE; Frédéric MERCIER, Pr, Study Chair — Hôpital Antoine Béclère - 92140 CLAMART; Alexandre MIGNON, Pr, Study Chair — Hôpital Cochin - 75014 PARIS; Cyril HUISSOUD, Pr, Study Chair — Hôpital Croix Rousse - 69004 LYON; Jean-Marie GROUIN, Study Chair — Université de Rouen - 76100 ROUEN
Locations (31):
- France (30):
  - CH Félix Guyon, Saint-Denis, Réunion
  - Groupe Hospitalier Sud Réunion, Saint-Pierre, Réunion
  - CHU d'Angers, Angers
  - Hôpital Privé d'Antony, Antony
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - Hôpital Femme Mère Enfant, Bron
  - Hôpital Antoine Béclère, Clamart
  - CHU Estaing, Clermont-Ferrand
  - Hôpital Louis Mourier, Colombes
  - Les Hôpitaux de Chartres (Hôpital Pasteur), Le Coudray
  - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Centre Hospitalier de Lens, Lens
  - CHU de Lille, Maternité Jeanne de Flandre, Lille
  - CHU de Limoges, Limoges
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Saint-Joseph / Pôle Parents - Enfants, Marseille
  - CHRU de Montpellier, Montpellier
  - Maternité Régionale Universitaire de Nancy, Nancy
  - Hôpital Necker - Enfants malades, Paris
  - Hôpital Armand Trousseau, Paris
  - Hôpital Cochin, Paris
  - Hôpital Tenon, Paris
  - CHU de Reims, Hôpital Maison Blanche, Reims
  - CHU de Rennes - Hôpital Sud, Rennes
  - Polyclinique de l'Atlantique, Saint-Herblain
  - Hôpital de Hautepierre, Strasbourg
  - Hôpital Foch, Suresnes
  - Hôpital Paul de Viguier - Site Purpan, Toulouse
  - CHU de Tours, Tours
  - CH de Valenciennes, Valenciennes
- CHR de Martinique, Fort-de-France, Martinique

REFERENCES:
- [Derived] Ducloy-Bouthors AS, Mercier FJ, Grouin JM, Bayoumeu F, Corouge J, Le Gouez A, Rackelboom T, Broisin F, Vial F, Luzi A, Capronnier O, Huissoud C, Mignon A; FIDEL working group. Early and systematic administration of fibrinogen concentrate in postpartum haemorrhage following vaginal delivery: the FIDEL randomised controlled trial. BJOG. 2021 Oct;128(11):1814-1823. doi: 10.1111/1471-0528.16699. Epub 2021 Apr 7. PMID 33713384

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between 10 April 2014 and 20 June 2018, 448 patients from 30 sites signed an informed consent.
Pre-assignment Details: During the pre-assigment period 11 patients withdrawn before treatment period. (1 treated with another IMP, 5 not treated, 2 no emergency consent signed, 1 no post inclusion consent signed, 2 refused to continue the study)
Groups:
- Clottafact: Human fibrinogen concentrate 3g intravenous use. 2 vials of 1,5 g/100mL, each vial of powder was reconstituted with 100 mL of sterile water for injection.
- Placebo: Placebo intravenous use. 2 vials of 100 mL, each vial of powder was reconstituted with 100 mL of sterile water.
Period: Treatment Period
Arm/Group | Clottafact | Placebo
Started | 224 | 213
Completed | 224 | 213
Not Completed | 0 | 0
Period: Follow-up Period
Arm/Group | Clottafact | Placebo
Started | 224 | 213
Completed | 207 | 202
Not Completed | 17 | 11

BASELINE CHARACTERISTICS:
Groups:
- Clottafact: Human fibrinogen concentrate 3g intravenous use. 2 vials of 1,5 g/100mL, each vial of powder was reconstitued with 100 mL of sterile water for injection.
- Placebo: Placebo intravenous use. 2 vials of 100 mL, eache vial of powder was reconttitued with 100 mL of sterile water for injection.
- Total: Total of all reporting groups
Arm/Group | Clottafact | Placebo | Total
Number analyzed (Participants) | 224 | 213 | 437
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 224 | 213 | 437
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (5.6) | 30.3 (5.4) | 30.4 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 224 | 213 | 437
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Failure Rate of PPH Management
Description: The primary efficacy variable is a binary (Failure versus Success) composite endpoint.
  Failure is defined when a patient:
  * loses at least 4 g/dL of Hb compared to the reference Hb level , AND/OR
  * requires the transfusion of at least 2 units of packed RBCs.
Time Frame: Evaluation of the two criteria that form the primary endpoint within the 48 h following the administration
Population: Number of patients with failure
Measure: Count of Participants; unit: Participants
Groups:
- Per Protocole (PP) Set Clottafact; Per Protocole (PP) Set Placebo: Patients with no missing data for the primary criterion.
- Intention To Treat (ITT) Set Clottafact: All patients treated with Clottafact. (patients who received at least one infusion of Clottafact)
- Intention To Treat (ITT) Set Placebo: All patients treated with Placebo. (patients who received at least one infusion of placebo)
- Full Analysis Set (FAS) Clottafact: Patients treated with Clottafact of the ITT Set with no missing data for the primary criteria.
- Full Analysis Set (FAS) Placebo: Patients treated with Placebo of the ITT Set with no missing data for the primary criteria.
Arm/Group | Per Protocole (PP) Set Clottafact | Per Protocole (PP) Set Placebo | Intention To Treat (ITT) Set Clottafact | Intention To Treat (ITT) Set Placebo | Full Analysis Set (FAS) Clottafact | Full Analysis Set (FAS) Placebo
Number analyzed (Participants) | 195 | 193 | 224 | 213 | 220 | 210
Participants | 75 | 80 | 92 | 92 | 88 | 89
Statistical Analysis 1: Comparison: Full Analysis Set (FAS) Clottafact vs Full Analysis Set (FAS) Placebo; Test type: Superiority; p = 0.9563, Regression, Logistic; Odds Ratio (OR) = 0.9889, 95% CI 2-sided [0.6633 to 1.4744]

2. Secondary Outcome: Patients With at Least Administration of 2 Units of RBCs
Description: Considering failure as the fact of requiring at least 2 units of RBCs.
Time Frame: from H0 to Day 2
Measure: Count of Participants; unit: Participants
Groups:
- FAS Set Clottafact: Patients treated with Clottafact of the ITT Set with no missing data for the primary criteria.
- FAS Set Placebo: Patients treated with Placebo of the ITT Set with no missing data for the primary criteria.
Arm/Group | FAS Set Clottafact | FAS Set Placebo
Number analyzed (Participants) | 220 | 210
Participants | 51 | 52
Statistical Analysis 1: Comparison: FAS Set Clottafact vs FAS Set Placebo; Failure on individual component of the primary endpoint defined as administration of 2 units of RBCs; Test type: Superiority; p = 0.9786, Regression, Logistic; Odds Ratio (OR) = 1.0064, 95% CI 2-sided [0.6321 to 1.6022]

3. Secondary Outcome: Patients With Loss of at Least 4 g/dL of Hb
Description: Considering failure as the fact of having lost at least 4 g/dL of Hb.
Time Frame: From reference value to Day 2
Measure: Count of Participants; unit: Participants
Arm/Group | FAS Set Clottafact | FAS Set Placebo
Number analyzed (Participants) | 220 | 210
Participants | 42 | 41
Statistical Analysis 1: Comparison: FAS Set Clottafact vs FAS Set Placebo; Failure on individual component of the primary endpoint defined as a loss of at least 4 g/dL of Hb; Test type: Superiority; p = 0.9474, Regression, Logistic; Odds Ratio (OR) = 1.0169, 95% CI 2-sided [0.6177 to 1.6741]

ADVERSE EVENTS:
Time Frame: The safety was assessed by recording all AEs occurring during the study, from signature of the informed consent to last study visit (6 +/- 2 weeks after delivery).
Groups:
- Placebo: Placebo intravenous use. 2 vials of 100 mL, eache vial of powder was reconttitued with 100 mL of sterile water.
Arm/Group | Clottafact | Placebo
All-Cause Mortality (participants affected / at risk) | 0/224 | 0/213
Serious Adverse Events (participants affected / at risk) | 10/224 | 10/213
Other Adverse Events (participants affected / at risk) | 95/224 | 106/213
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clottafact (N=224) | Placebo (N=213)
Aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Blood pressure inadequately controlled (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Shock haemorrhagic (Vascular disorders) | 1 (1) | 0 (0)
Thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1)
Blood pressure ambulatory increased (Investigations) | 1 (1) | 0 (0)
Blood uric acid increased (Investigations) | 0 (0) | 1 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (1)
HELLP syndrome (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Retained placenta or membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 1 (1)
Discomfort (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Psychological trauma (Psychiatric disorders) | 1 (1) | 0 (0)
Broad ligament haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Metrorrhagia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Uterine necrosis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine rupture (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute fatty liver of pregnancy (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Amniotic cavity infection (Infections and infestations) | 1 (1) | 0 (0)
Endometritis decidual (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis acute (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clottafact (N=224) | Placebo (N=213)
Hypertension (Vascular disorders) | 3 (3) | 6 (6)
Hypotension (Vascular disorders) | 5 (5) | 4 (4)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3)
Headache (Nervous system disorders) | 5 (6) | 7 (8)
Hyperthermia (General disorders) | 2 (2) | 5 (5)
Influenza like illness (General disorders) | 0 (0) | 3 (3)
Oedema peripheral (General disorders) | 4 (4) | 6 (6)
Pyrexia (General disorders) | 11 (11) | 12 (12)
Malaise (General disorders) | 2 (2) | 4 (4)
Anxiety (Psychiatric disorders) | 3 (3) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 1 (1)
Constipation (Gastrointestinal disorders) | 9 (9) | 4 (4)
Haemorrhoids (Gastrointestinal disorders) | 21 (21) | 29 (29)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 1 (1) | 4 (4)
Metrorrhagia (Reproductive system and breast disorders) | 6 (6) | 3 (3)
Nipple disorder (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Oedema genital (Reproductive system and breast disorders) | 2 (2) | 5 (5)
Uterine pain (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Vulval oedema (Reproductive system and breast disorders) | 0 (0) | 4 (4)
Hepatocellular injury (Hepatobiliary disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Endometritis decidual (Infections and infestations) | 4 (4) | 5 (5)
Puerperal pyrexia (Infections and infestations) | 7 (7) | 4 (4)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (3):
  • Study Protocol (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT02155725/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/25/NCT02155725/SAP_001.pdf
  • Informed Consent Form (2018-03-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT02155725/ICF_002.pdf